CLINICAL TRIAL: NCT06626724
Title: A Retrospective Cohort Study on Predicting Delayed Graft Function in Liver Transplant Patients with Hepatocellular Carcinoma: a Nomogram and Machine Learning Approaches.
Status: Completed | Type: Observational
Sponsor: Jian You (Other)
Responsible Party: Sponsor-Investigator, Jian You, Research assistant, Wuhan University
Organization: Wuhan University (Other)
Other Study IDs: Zhongnan Hospital
Record Dates: First submitted 2024-10-01; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma (HCC); DGF
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Liver transplantation — Liver transplantation for patients with hepatocellular carcinoma.

SUMMARY:
Background: This study aimed to develop a predictive model for delayed graft function (DGF) in liver transplant patients with hepatocellular carcinoma (HCC) based on preoperative biochemical indicators, using both logistic regression and XGBoost machine learning algorithms.

Methods: A retrospective cohort study was conducted, including 131 liver transplant patients from January 2020 to April 2022. Preoperative biochemical markers and hematological parameters were analyzed. Logistic regression and XGBoost models were constructed to predict DGF, and their performance was evaluated using the area under the ROC curve (AUC). Shapley Additive Explanations (SHAP) analysis was employed to interpret the feature contributions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with liver cancer aged between 18 and 75 years.
2. Patients who have received liver transplantation.
3. Complete preoperative and postoperative medical imaging data, clinical records and pathological test reports are available.

Exclusion Criteria:

1. Primary non-hepatocellular carcinoma
2. Recipients were younger than 18 years and older than 75 years
3. Due to incomplete or missing clinical data, this dataset did not meet the criteria for inclusion in the statistical analysis.
4. Serious complications associated with liver transplantation, such as acute transplant rejection or transplant liver failure, occur within 7 days after surgery.
5. Re-surgery within 7 days after surgery due to liver transplant-related complications or other surgical procedures, such as transplant site infection or other major surgery.

Ages: 18 Days to 75 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients receiving a liver transplant between January 2020 and April 2024.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
TBIL/AST/ALT/INR | Results of biochemical examination on the 7th day after liver transplantation in patients with hepatocellular carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The data are not publicly available, as participants in this study need their data for further analysis.